CLINICAL TRIAL: NCT07283861
Title: A Phase 2 Trial of Accessory Nerve Wrapping With the Axoguard HA Plus Nerve Protector to Reduce Post-operative Neck and Shoulder Dysfunction in Patients Undergoing Neck Dissection
Brief Title: Axoguard HA Plus Nerve Protector to Reduce Post-operative Neck and Shoulder Dysfunction in Patients Undergoing Neck Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Spector (Other)
Collaborators: Axogen Corporation (Industry)
Responsible Party: Sponsor-Investigator, Matthew Spector, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25060040
Record Dates: First submitted 2025-12-06; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Neck Dissection
Keywords: shoulder function; neck dissection; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Axoguard HA+ Arm (Experimental)
  Interventions: Device: Spinal Accessory Nerve Protection utilizing Axoguard HA+

INTERVENTIONS:
Device: Spinal Accessory Nerve Protection utilizing Axoguard HA+ — Nerve protection utilizing a nerve wrap.

SUMMARY:
In this prospective study, patients with head and neck cancers undergoing neck dissection will have the nerve to the shoulder wrapped with the Axoguard HA+ Nerve Protector at time of surgery. In these patients, the presence and severity of neck and shoulder dysfunction on the operated side will be assessed approximately twelve months post-operatively. The investigators hypothesize that shoulder nerve wrapping with the Axoguard HA+ Nerve Protector will lead to clinically meaningful improvement of shoulder function.

DETAILED DESCRIPTION:
All patients will undergo neck dissection and the spinal accessory nerve wrapped with the Axoguard HA+ Nerve Protector. The Neck Dissection Impairment Index will be administered before surgery and 1 year after surgery and compared to historical controls. The NDII is on a 100 point scale with a higher score indicating a better shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated malignancy of the head and neck including primary mucosal, cutaneous, salivary gland, and thyroid cancers
* Undergoing accessory-nerve sparing elective or therapeutic SND or MRND (involving level II and/or level V dissection)
* 18 years or older
* Patients must give documented informed consent to participate in this study

Exclusion Criteria:

* Previous history of neck or shoulder surgery or radiation
* Inadvertent injury to or intentional sacrifice of the accessory nerve at time of neck dissection
* Medical contraindication to surgery under general anesthesia
* Known sensitivity to porcine materials
* Pregnant or lactating patients
* Incarcerated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
One year neck and shoulder dysfunction as assessed by the neck dissection impairment index | one year
  The neck dissection impairment index is a score from 1-100 with 100 being a perfect score.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zandberg, Study Chair — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12-1-25 to completion of study
Access Criteria: Available upon request